CLINICAL TRIAL: NCT07019051
Title: Predictive Role of Echocardiographic Parameters for Hemodynamic Support Needs During Initiation of Continuous Venovenous Hemodiafiltration in ICU Patients
Brief Title: Echocardiographic Parameters for Hemodynamic Support During CVVHDF
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: lvot vti AKIN
Record Dates: First submitted 2025-05-28; First posted 2025-06-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CVVHDF Candidates in ICU: Adult intensive care unit (ICU) patients who are scheduled to undergo continuous veno-venous hemodiafiltration (CVVHDF). All participants will undergo transthoracic echocardiographic evaluation prior to dialysis initiation. Hemodynamic parameters will be monitored for 60 minutes following the start of CVVHDF to assess the development of hypotension or the need for vasopressor, inotropic, or fluid support.
  Interventions: Diagnostic Test: Transthoracic Echocardiographic Evaluation

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiographic Evaluation — Non-invasive transthoracic echocardiography will be performed prior to the initiation of continuous veno-venous hemodiafiltration (CVVHDF) in ICU patients. The evaluation includes measurements of LVOT VTI, MAPSE, TAPSE, S' wave velocity, and E/e' ratio to assess cardiac function and estimate the risk of hemodynamic instability. The procedure will be conducted at the bedside using standard parasternal and apical windows by trained intensive care physicians or cardiologists. No contrast, sedation, or invasive monitoring will be used.

SUMMARY:
This prospective observational study aims to evaluate whether transthoracic echocardiographic parameters-Left Ventricular Outflow Tract Velocity-Time Integral (LVOT VTI), Mitral Annular Plane Systolic Excursion (MAPSE), Tricuspid Annular Plane Systolic Excursion (TAPSE), S' wave velocity, and E/e' ratio-can predict hemodynamic instability at the initiation of sustained low-efficiency daily dialysis (SVVHDF) in intensive care unit (ICU) patients. The study will include adult patients requiring SVVHDF, and echocardiographic measurements will be performed prior to dialysis. The primary outcome is the need for hemodynamic support (vasopressors/inotropes or fluid resuscitation) or development of hypotension within the first 60 minutes of dialysis. The study aims to identify which of these parameters best predict the need for hemodynamic intervention, with the goal of supporting individualized dialysis planning and safer fluid management in critically ill patients.

DETAILED DESCRIPTION:
This prospective, single-center observational study is designed to investigate the predictive value of specific transthoracic echocardiographic (TTE) parameters in assessing the risk of hemodynamic instability during the initiation of sustained low-efficiency daily dialysis (SVVHDF) in critically ill patients. The primary focus is to determine whether measurements obtained immediately before dialysis-namely LVOT VTI, MAPSE, TAPSE, S', and E/e'-can identify patients at risk of hypotension or the need for hemodynamic support within the first hour of treatment.

All echocardiographic assessments will be performed by certified intensive care specialists or cardiologists using standard parasternal and apical windows. The parameters to be evaluated include:

LVOT VTI (Left Ventricular Outflow Tract Velocity-Time Integral):

Measured via pulsed wave Doppler from the apical 5-chamber view, this value reflects stroke volume and overall cardiac output. A low LVOT VTI may indicate hypovolemia or decreased systolic function.

MAPSE (Mitral Annular Plane Systolic Excursion):

Obtained using M-mode in the apical 4-chamber view by measuring the displacement of the mitral annulus during systole. It is an index of longitudinal left ventricular systolic function; values <10 mm may suggest early left ventricular dysfunction.

TAPSE (Tricuspid Annular Plane Systolic Excursion):

Also measured with M-mode in the apical 4-chamber view, TAPSE reflects right ventricular systolic function. Values <17 mm are indicative of right ventricular dysfunction.

S' (S Prime) Wave:

Using tissue Doppler imaging (TDI) at the mitral and/or tricuspid annulus, this parameter evaluates longitudinal systolic myocardial velocity. Reduced S' values suggest impaired ventricular contractility.

E/e' Ratio:

Calculated from pulsed Doppler and TDI values, this ratio estimates left ventricular filling pressures. An E/e' >15 is associated with elevated filling pressure, while <8 suggests normal filling.

Patients will be monitored for hemodynamic instability within the first 60 minutes following SVVHDF initiation. The primary hemodynamic outcomes include:

Hypotension: Defined as a mean arterial pressure (MAP) <65 mmHg or a ≥20% decrease in MAP compared to baseline values prior to dialysis initiation.

Need for Vasopressor or Inotrope Support: Initiation of medications such as norepinephrine, dopamine, or dobutamine during the first hour of dialysis.

Need for Additional Fluid Resuscitation: Defined as administration of ≥500 mL crystalloid or colloid solution within 60 minutes due to clinical signs of volume depletion.

Clinical decisions related to dialysis and hemodynamic management will be made solely by the treating physicians, with study investigators collecting data in an observational capacity. All echocardiographic and hemodynamic data will be anonymized and stored securely for statistical analysis.

This study aims to identify echocardiographic biomarkers that can improve the safety and personalization of dialysis management in ICU settings, with potential applications extending to chronic dialysis centers in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Admission to the intensive care unit (ICU)
* Clinical indication for initiation of continuous veno-venous hemodiafiltration (CVVHDF)
* Ability to obtain adequate transthoracic echocardiographic (TTE) images prior to CVVHDF
* Written informed consent obtained from the patient's legal representative

Exclusion Criteria:

* Acute coronary syndrome, severe valvular disease, or pericardial effusion affecting cardiac function
* Cardiac arrhythmias such as atrial fibrillation or ventricular tachycardia that interfere with accurate Doppler measurements
* Presence of cardiac devices such as pacemakers, LVADs, or implantable cardioverter defibrillators (ICDs)
* Poor echocardiographic window due to severe lung disease or chest wall abnormalities
* Estimated life expectancy <24 hours or do-not-resuscitate (DNR) orders in place
* Inability to obtain informed consent due to lack of legal representative
* Transfer to another facility before CVVHDF initiation or change in renal replacement strategy (e.g., switch to peritoneal dialysis)
* Incomplete echocardiographic measurement due to technical limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years) admitted to the intensive care unit (ICU) of a tertiary care hospital who are clinically indicated for continuous veno-venous hemodiafiltration (CVVHDF) due to acute kidney injury or fluid overload. All participants must have adequate transthoracic echocardiographic imaging quality prior to dialysis initiation. Only patients whose legal representatives provide informed consent will be included. Both male and female patients will be enrolled, regardless of underlying comorbidities, provided they meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of Hemodynamic Instability Within the First 60 Minutes of CVVHDF and Its Association With Pre-Dialysis LVOT VTI | Within the first 60 minutes of CVVHDF initiation
  Hemodynamic instability will be recorded within the first 60 minutes after initiation of continuous veno-venous hemodiafiltration (CVVHDF). Instability is defined by the occurrence of any of the following:
  Mean arterial pressure (MAP) < 65 mmHg,
  ≥30% decrease in MAP from pre-CVVHDF baseline,
  Initiation of vasopressors or inotropes,
  Administration of ≥500 mL of intravenous fluid bolus for resuscitation.
  Each patient's Left Ventricular Outflow Tract Velocity-Time Integral (LVOT VTI) will be measured by transthoracic echocardiography prior to CVVHDF initiation.

SECONDARY OUTCOMES:
Association Between Pre-Dialysis MAPSE Values and Hemodynamic Instability Within the First 60 Minutes of CVVHDF | Within the first 60 minutes of CVVHDF initiation
  Mitral Annular Plane Systolic Excursion (MAPSE) will be measured using transthoracic echocardiography prior to the initiation of continuous veno-venous hemodiafiltration (CVVHDF). Hemodynamic instability will be defined as the occurrence of any of the following events within 60 minutes of CVVHDF initiation:
  Mean arterial pressure (MAP) < 65 mmHg,
  ≥30% reduction in MAP from baseline,
  Need for vasopressors or inotropes,
  Requirement of ≥500 mL intravenous fluid bolus.
Association Between Pre-Dialysis TAPSE Values and Hemodynamic Instability Within the First 60 Minutes of CVVHDF | Within the first 60 minutes of CVVHDF initiation
  Tricuspid Annular Plane Systolic Excursion (TAPSE) will be measured using transthoracic echocardiography prior to the initiation of continuous veno-venous hemodiafiltration (CVVHDF). Hemodynamic instability will be recorded during the first 60 minutes after CVVHDF initiation and defined as the occurrence of any of the following:
  Mean arterial pressure (MAP) < 65 mmHg,
  ≥30% reduction in MAP from baseline,
  Use of vasopressors or inotropes,
  Administration of ≥500 mL of intravenous fluid for resuscitation.
Association Between Pre-Dialysis S' Wave Velocity (cm/s) Measured by Tissue Doppler Imaging and Hemodynamic Instability During the First 60 Minutes of CVVHDF | Within the first 60 minutes of CVVHDF initiation
  Systolic S' wave velocity (in cm/s) will be measured by tissue Doppler imaging of the tricuspid annulus via transthoracic echocardiography prior to the initiation of continuous veno-venous hemodiafiltration (CVVHDF). Hemodynamic instability will be defined as any of the following occurring within the first 60 minutes of dialysis:
  Mean arterial pressure (MAP) < 65 mmHg,
  ≥30% decrease in MAP from baseline,
  Requirement for vasopressors or inotropes,
  Administration of ≥500 mL intravenous fluid bolus.
Association Between Pre-Dialysis E/e' Ratio and Hemodynamic Instability Within the First 60 Minutes of CVVHDF | Within the first 60 minutes of CVVHDF initiation
  The E/e' ratio will be calculated using pulsed-wave Doppler (for mitral inflow E wave) and tissue Doppler imaging (for early diastolic mitral annular e' velocity) obtained via transthoracic echocardiography prior to initiation of continuous veno-venous hemodiafiltration (CVVHDF).
  Hemodynamic instability will be defined as the occurrence of any of the following within the first 60 minutes of CVVHDF:
  Mean arterial pressure (MAP) < 65 mmHg,
  ≥30% decrease in MAP from baseline,
  Initiation of vasopressors or inotropes,
  Requirement for ≥500 mL intravenous fluid bolus.

CONTACTS AND LOCATIONS:
Overall Officials: Engin ihsan Turan, Specialist, Principal Investigator — Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to qualified researchers upon reasonable request. The shared data will include echocardiographic parameters (LVOT VTI, MAPSE, TAPSE, S', E/e'), hemodynamic measurements, and outcome data related to the development of hemodynamic instability following the initiation of CVVHDF. Personal identifiers will be removed to ensure privacy and compliance with ethical standards.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD and supporting materials will be available beginning 6 months after the publication of the study results and will remain available for 1 years.
Access Criteria: Access to data will be granted to researchers who provide a methodologically sound research proposal, approved by an independent review committee. Requests should be submitted to the principal investigator. A data-sharing agreement outlining the terms of use, data protection, and intended analyses will be required prior to data release.